CLINICAL TRIAL: NCT04513028
Title: Beta Glucan's Effect on Pembrolizumab Immunologic Response in Stage III-IV Melanoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kelly McMasters (Other)
Responsible Party: Sponsor-Investigator, Kelly McMasters, Principal Investigator, University of Louisville
Organization: University of Louisville (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20.0614
Record Dates: First submitted 2020-07-30; First posted 2020-08-14 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Melanoma Stage III; Melanoma Stage IV
MeSH Terms: conditions — Melanoma | interventions — beta-Glucans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All subjects will undergo 21 days of Pembrolizumab followed by 21 days of beta-glucan.
  Pembrolizumab: 200 mg/100mL IV in three week intervals
  Beta-glucan: 500mg (1 capsule) by mouth twice a day for 21 days
  Interventions: Dietary Supplement: Beta-Glucan

INTERVENTIONS:
Dietary Supplement: Beta-Glucan — 500mg (1 capsule) by mouth twice a day for 21 days.

SUMMARY:
The purpose of this study is to determine how beta-glucan affects the immune system in subjects with melanoma.

DETAILED DESCRIPTION:
This is a clinical pilot study using oral beta-glucan on patients with advanced stage III-IV melanoma without evidence of disease receiving adjuvant Pembrolizumab. The aim is to see whether beta-glucan treatment in combination with Pembrolizumab may provide augmented immunologic phenotypes such as decreased peripheral MDSCs, enhanced T effector cell function, or enhanced cytokine production in the peripheral blood or plasm of enrolled subjects. Secondary outcome measures will include clinical endpoints such as recurrence, progression free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Any patients with suspected (clinical) or definitive (tissue) diagnosis of Stage III-IV melanoma starting or continuing adjuvant Pembrolizumab without active evidence of disease (NED).
* Must be treatment naïve or have had treatment no less than 6 months prior to enrollment
* 18 years or older
* Must be able to take pills
* ECOG performance status of 0-3
* Ability to understand and willingness to sign a written informed consent
* Members of all racial and ethnic groups are eligible for this study

Exclusion Criteria:

* History of hypersensitivity reactions attributed to beta-glucan
* Patients receiving continuous or other ongoing immunosuppressive therapy
* Uncontrolled intercurrent illness including, but not limited to, autoimmune diseases, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any patients who have serious autoimmune toxicity during the study period, or those who have disease recurrence during the 6-week study period should be excluded and analyzed separately
* Patients with mucosal melanoma
* Patients with concurrent malignancy or recent history thereof

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Changes in percent of lymphocyte cell surface expression markers | Blood for analysis will be drawn at baseline (Day 0), 3 weeks post pembrolizumab treatment, and 3 weeks post pembrolizumab plus oral beta-glucan treatment.
  The investigators will quantify percent of lymphocyte cell surface e (i.e., CD45, CD3, CD11b, etc.) from each sample collected by mass cytometry *CyTOF) or flow cytometry
Changes in absolute number of lymphocyte cell surface expression markers | Blood for analysis will be drawn at baseline (Day 0), 3 weeks post pembrolizumab treatment, and 3 weeks post pembrolizumab plus oral beta-glucan
  The investigators will quantify absolute number of lymphocyte cell surface (i.e., CD45, CD3, CD11b, etc.) from each sample collected by mass cytometry (CyTOF) or flow cytometry
Changes in the mean fluorescent intensity of lymphocyte cell surface expression markers | Blood for analysis will be drawn at baseline (Day 0), 3 weeks post pembrolizumab treatment, and 3 weeks post pembrolizumab plus oral beta-glucan
  The investigators will quantify mean fluorescent intensity of lymphocyte cell surface (i.e., CD45, CD3, CD11b, etc.) from each sample collected by mass cytometry *CyTOF) or flow cytometry
Changes in percent of intracellular cytokine expression markers | Blood for analysis will be drawn at baseline (Day 0), 3 weeks post pembrolizumab treatment, and 3 weeks post pembrolizumab plus oral beta-glucan
  The investigators will quantify percent of intracellular cytokine expression (TNFa, IFNg, etc.) from each sample collected by mass cytometry (CyTOF) or flow cytometry
Changes in absolute number of intracellular cytokine expression markers | Blood for analysis will be drawn at baseline (Day 0), 3 weeks post pembrolizumab treatment, and 3 weeks post pembrolizumab plus oral beta-glucan
  The investigators will quantify absolute number of intracellular cytokine expression (TNF-a, IFNg, etc.) from each sample collected by mass cytometry (CyTOF) or flow cytometry
Changes in fluorescent intensity of intracellular cytokine expression markers | Blood for analysis will be drawn at baseline (Day 0), 3 weeks post pembrolizumab treatment, and 3 weeks post pembrolizumab plus oral beta-glucan
  The investigators will quantify fluorescent intensity of intracellular cytokine expression (TNF-a, IFNg, etc.) from each sample collected by mass cytometry (CyTOF) or flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Kelly M McMasters, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No